CLINICAL TRIAL: NCT03035864
Title: A 8 Weeks, Phase II, Single-centre, Randomized, Double-masked, Vehicle-controlled, Parallel Group Study With 4 Weeks Follow-up to Evaluate Efficacy & Safety of rhNGF Eye Drops vs Vehicle in Patients After Cataract and Refractive Surgery
Brief Title: A 8 Weeks Study to Evaluate Efficacy & Safety of rhNGF vs Vehicle in Patients After Cataract and Refractive Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NGF0116
Record Dates: First submitted 2017-01-23; First posted 2017-01-30 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-12

CONDITIONS: Ocular Discomfort
Keywords: Ocular discomfort after cataract and refractive surgery; cataract surgery; refractive surgery
MeSH Terms: interventions — Nerve Growth Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: For the whole duration of the trial, treatment was unknown to the patient, the Investigator and the site staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhNGF 20 µg/ml (Experimental): Recombinant Human Nerve Growth Factor (rhNGF) at 20 μg/mL eye drops six times daily
  Interventions: Drug: rhNGF
- Vehicle (Placebo Comparator): Vehicle eye drops six times daily
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: rhNGF — Eye Drop 20 μg/mL
  Other Names: NGF
  Arms: rhNGF 20 µg/ml
Other: Vehicle — Vehicle Eye Drop
  Arms: Vehicle

SUMMARY:
The primary objective of this exploratory study is to assess preliminary efficacy and safety of rhNGF when administered as eye drops to patients after cataract and refractive surgery.

The main criteria for evaluation were:

* Change from baseline in SANDE scores for severity and frequency assessed at 8 weeks of treatment (primary efficacy endpoint)
* Changes in Cornea vital staining with fluorescein (National Eye Institute [NEI] scales) assessed at 8 weeks of treatment (co-primary efficacy endpoint)
* Changes in conjunctiva vital staining with fluorescein (NEI scales) (secondary efficacy endpoint);
* Changes in Tear Film Break-Up Time (TFBUT)(secondary efficacy endpoint);
* Changes in Cochet-Bonnet corneal aesthesiometry (secondary efficacy endpoint);
* Changes in Nerve count and morphology at scanning laser in vivo corneal confocal microscopy (only patients who had Laser-Assisted In situ Keratomileusis [LASIK] surgery) (secondary efficacy endpoint);
* Changes in SANDE scores (face values) for severity and frequency (secondary efficacy endpoint);
* Incidence and frequency of treatment-emergent adverse events (TEAEs), assessed throughout the study (safety endpoint).

DETAILED DESCRIPTION:
The proposed phase II study is a single-centre, randomized, double masked, parallel arm, vehicle-controlled trial, designed to evaluate the preliminary efficacy and safety of rhNGF eye drops at 20 µg/ml concentration administered six times daily for 8 weeks in patients who underwent cataract and corneal refractive surgery, both known to damage the corneal sensory nerve plexus.

After confirmation of inclusion and exclusion criteria all eligible patients will be randomized at 2:1 ratio to rhNGF or vehicle control treatment with 8 weeks of study treatments administration with 4 weeks Follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years old
2. Patients who are characterized by the following clinical features:

   1. History of cataract or refractive corneal surgery in the study eye(s) in the previous 6 months;
   2. Mean Symptom Assessment in Dry Eye (SANDE) score for severity and frequency of at least 30 at baseline
3. The same eye (study eye) must fulfill all the above criteria
4. Best corrected distance visual acuity (BCDVA) score of ≥ 0.1 decimal units in both eyes at the time of study enrolment
5. Female patients must have negative pregnancy urine test if at childbirth potential.
6. Only patients who satisfy all requirements for informed consent may be included in the study. Written Informed Consent must be obtained before the initiation of any study-specific procedures.
7. Patients must have the ability and willingness to comply with study procedures

Exclusion Criteria:

1. Any ocular disease other than Dry Eye requiring treatment with topical medications in either eye at the time of study enrolment.
2. Any active ocular infection or active inflammation in either eye unrelated to Dry Eye.
3. Presence or history of any systemic or ocular disorder, condition or disease (with particular attention to malignancies and neuro-oncological diseases) that could possibly interfere with the conduct of the required study procedures or the interpretation of the study results.
4. Use of therapeutic or Refractive Contact lenses in either eye at the time of study enrolment;
5. History of ocular surgery in the study eye(s), excluding corneal refractive or cataract procedures, within 90 days of study enrolment.
6. Females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) are excluded from participation in the study if they meet any one of the following conditions:

   1. are currently pregnant or,
   2. have a positive result at the urine pregnancy test (Baseline/Day 0) or,
   3. intend to become pregnant during the study treatment period or,
   4. are breast-feeding or,
   5. are not willing to use highly effective birth control measures, such as: hormonal contraceptives - oral, implanted, transdermal, or injected - and/or mechanical barrier methods - spermicide in conjunction with a barrier such as a condom or diaphragm or IUD (Intrauterine device) - during the entire course of and 30 days after the study treatment periods.
7. Participation in another clinical study at the same time as the present and within 30 days of study enrolment;
8. History of drug, medication or alcohol abuse or addiction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Mastropasqua, MD, Principal Investigator — Univ. G. D'Annunzio- Clinica Oftalmologica Chieti
Locations (1):
- Univ. G. D'Annunzio-Clinica Oftalmologica-Chieti, Chieti, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were randomized in a 2:1 ratio to rhNGF eye drops solution at 20 μg/ml (120 patients) or vehicle eye drops solution (60 patients) 6 times per day for 8 weeks, followed by 4 weeks of follow-up with no further treatment.
Period: Treatment Period
Arm/Group | rhNGF 20 µg/ml | Vehicle
Started | 120 | 60
Completed | 116 | 59
Not Completed | 4 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Other | 3 | 1
Period: Follow-up Period
Arm/Group | rhNGF 20 µg/ml | Vehicle
Started | 116 | 59
Completed | 105 | 55
Not Completed | 11 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 6 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Other | 3 | 2

BASELINE CHARACTERISTICS:
Population: Analysed for safety (SAF) population
Groups:
- Total: Total of all reporting groups
Arm/Group | rhNGF 20 µg/ml | Vehicle | Total
Number analyzed (Participants) | 115 | 59 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (12.80) | 34.4 (11.20) | 36.8 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 33 | 104
  Male | 44 | 26 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 115 | 57 | 172
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 115 | 59 | 174

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in SANDE Scores for Frequency and Severity Assessed at 8 Weeks of Treatment.
Description: The Symptom Assessment in Dry Eye (SANDE) questionnaire is a short questionnaire to evaluate both dry eye intensity and frequency by using a 100 mm visual analogue scale (VAS). The patient symptoms of ocular dryness and/or irritation were quantified on the scale based on two questions that assessed both the severity and frequency of symptoms.
  The SANDE score is calculated by taking the square root of the product of the frequency of symptoms score and the severity of symptoms score. The SANDE scale ranges from 0 to 100 with 100 being the maximal amount of dry eye symptoms and 0 being the minimal amount of dry eye symptoms.
Time Frame: Baseline and Week 8
Population: Full Analysis Set Population. Last observation carried forward (LOCF) imputation method
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF 20 µg/ml | Vehicle
Number analyzed (Participants) | 112 | 58
score on a scale
  Frequency | -37.2 (24.85) | -35.7 (26.04)
  Severity | -37.8 (27.20) | -37.3 (20.43)
Statistical Analysis 1: Comparison: rhNGF 20 µg/ml vs Vehicle; Frequency statistical analysis; Test type: Superiority; p = 0.974, ANCOVA; difference in LS means = -0.11, 95% CI 2-sided [-6.85 to 6.63]
Statistical Analysis 2: Comparison: rhNGF 20 µg/ml vs Vehicle; Statistical analysis related to severity; Test type: Superiority; p = 0.399, ANCOVA; Difference in least square means = 2.88, 95% CI 2-sided [-3.85 to 9.61]

2. Primary Outcome: Changes in Cornea Vital Staining With Fluorescein (National Eye Institute [NEI] Scales)
Description: Corneal Staining was derived as the sum of scores of the five corneal sectors (central, superior, inferior, nasal, and temporal) each of which was scored on a scale of 0-3, with a minimum score of 0 and a maximal score of 15 (sum > 3 out of 15 is abnormal).
Time Frame: Baseline and Week 8
Population: Full Analysis Set population. Last observation carried forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF 20 µg/ml | Vehicle
Number analyzed (Participants) | 112 | 58
score on a scale | -2.5 (2.11) | -2.2 (1.81)
Statistical Analysis 1: Comparison: rhNGF 20 µg/ml vs Vehicle; Test type: Superiority; p = 0.214, ANCOVA; difference in least square means = 0.04, 95% CI 2-sided [-0.02 to 0.10]

3. Secondary Outcome: Changes in Conjunctiva Vital Staining With Fluorescein (National Eye Institute [NEI] Scales)
Description: Conjunctival Staining was derived as the sum of scores of the conjunctival area (nasal-superior paralimbal, nasal-inferior paralimbal, nasal-peripheral, temporal-superior paralimbal, temporal-inferior paralimbal, temporal-peripheral) with a grading scale of 0-3 and with a minimum score of 0 and a maximal score of 18 (18 indicates the most abnormal score). Grades increase with the number and density of dots.
  Data for the main eye are reported.
Time Frame: From baseline to weeks 4, 8 and 12
Population: As of this secondary endpoint, FAS Population was taken into account, but the last observation carried forward (LOCF) imputation method was not applied. Due to the reason mentioned above, the patients actually analysed (n) were the following:
  Week 4 - 110 rhNGF; 58 vehicle Week 8 - 107 rhNGF; 58 vehicle Week 12 - 107 rhNGF; 55 vehicle
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rhNGF 20 µg/ml | Vehicle
Number analyzed (Participants) | 112 | 58
units on a scale
  week 4: number analyzed (Participants) | 110 | 58
  week 4 | 0.0 (0.00) | 0.0 (0.00)
  week 8: number analyzed (Participants) | 107 | 58
  week 8 | 0.0 (0.00) | 0.0 (0.00)
  week 12: number analyzed (Participants) | 107 | 55
  week 12 | 0.0 (0.00) | 0.0 (0.00)

4. Secondary Outcome: Changes in Tear Film Break-Up Time (TFBUT)
Description: The TFBUT measurement was performed after instillation of 5 microliters of 2% sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye. The patient was instructed to blink several times to thoroughly mix the fluorescein with the tear film.
  Data for the main eye are reported.
Time Frame: From baseline to weeks 4, 8 and 12
Population: As of this secondary endpoint, FAS Population was taken into account, but the last observation carried forward (LOCF) imputation method was not applied. Due to the reason mentioned above, the patients actually analysed (n) were the following:
  Week 4 - 110 rhNGF Week 8 - 107 rhNGF Week 12 - 107 rhNGF
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | rhNGF 20 µg/ml | Vehicle
Number analyzed (Participants) | 112 | 58
seconds
  week 4: number analyzed (Participants) | 110 | 58
  week 4 | 2.5 (3.07) | 2.5 (2.37)
  week 8: number analyzed (Participants) | 107 | 58
  week 8 | 1.9 (2.96) | 2.2 (2.67)
  week 12: number analyzed (Participants) | 107 | 58
  week 12 | 2.3 (2.61) | 2.7 (2.72)

5. Secondary Outcome: Changes in Cochet-Bonnet Corneal Aesthesiometry
Description: Corneal sensation was measured in both eyes in each of the four quadrants of the cornea using the Cochet Bonnet aesthesiometer before the instillation of any dilating or anesthetic eye drops. The handheld esthesiometer (Cochet-Bonnet) is a device that contains a thin, retractable, nylon monofilament that extends up to 6 cm in length. Variable pressure can be applied by the device by adjusting the length. The monofilament ranges from 60 mm to 5 mm and as the length is decreased the pressure increases from 11 mm/gm to 200 mm/gm.
  Data for the main eye are reported.
Time Frame: From baseline to week 8
Population: As of this secondary endpoint, FAS Population was taken into account, but the last observation carried forward (LOCF) imputation method was not applied.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | rhNGF 20 µg/ml | Vehicle
Number analyzed (Participants) | 107 | 58
cm
  superior nasal | -0.1 (0.31) | -0.2 (0.31)
  inferior nasal | -0.2 (0.32) | -0.1 (0.64)
  superior temporal | -0.2 (0.36) | -0.2 (0.34)
  inferior temporal | -0.1 (0.41) | 0.0 (0.64)

6. Secondary Outcome: Changes in SANDE Scores (Face Values) for Frequency and Severity
Description: as for outcome 1
Time Frame: From baseline to weeks 4, 8 and 12
Population: Full Analysis Set Population. Observed values are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF 20 µg/ml | Vehicle
Number analyzed (Participants) | 112 | 58
score on a scale
  Frequency - week 4: number analyzed (Participants) | 110 | 58
  Frequency - week 4 | -35.1 (22.37) | -33.2 (25.18)
  Frequency - week 8: number analyzed (Participants) | 107 | 58
  Frequency - week 8 | -37.2 (24.84) | -35.7 (26.04)
  Frequency - week 12: number analyzed (Participants) | 107 | 55
  Frequency - week 12 | -42.1 (22.94) | -38.6 (26.25)
  Severity - week 4: number analyzed (Participants) | 110 | 58
  Severity - week 4 | -35.7 (24.28) | -32.9 (20.03)
  Severity - week 8: number analyzed (Participants) | 107 | 58
  Severity - week 8 | -37.9 (27.51) | -37.3 (20.43)
  Severity - week 12: number analyzed (Participants) | 107 | 55
  Severity - week 12 | -43.5 (22.7) | -38.4 (20.23)
Statistical Analysis 1: Comparison: rhNGF 20 µg/ml vs Vehicle; Frequency - week 4; Test type: Superiority; p = 0.881, ANCOVA; difference in least square means = -0.43, 95% CI 2-sided [-6.13 to 5.27]
Statistical Analysis 2: Comparison: rhNGF 20 µg/ml vs Vehicle; Frequency - week 8; Test type: Superiority; p = 0.926, ANCOVA; difference in least square means = -0.31, 95% CI 2-sided [-6.96 to 6.33]
Statistical Analysis 3: Comparison: rhNGF 20 µg/ml vs Vehicle; Frequency - Week 12; Test type: Superiority; p = 0.426, ANCOVA; difference in least square means = -2.29, 95% CI 2-sided [-7.97 to 3.38]
Statistical Analysis 4: Comparison: rhNGF 20 µg/ml vs Vehicle; Severity - Week 4; Test type: Superiority; p = 0.828, ANCOVA; Difference in least square means = 0.62, 95% CI 2-sided [-5.04 to 6.29]
Statistical Analysis 5: Comparison: rhNGF 20 µg/ml vs Vehicle; Severity - Week 8; Test type: Superiority; p = 0.394, ANCOVA; difference in least square means = 2.86, 95% CI 2-sided [-3.75 to 9.47]
Statistical Analysis 6: Comparison: rhNGF 20 µg/ml vs Vehicle; Severeity - Week 12; Test type: Superiority; p = 0.552, ANCOVA; difference in least square means = -1.49, 95% CI 2-sided [-6.41 to 3.44]

ADVERSE EVENTS:
Time Frame: Adverse events were collected at each time point of the study (ie. Baseline visit, Week 4, Week 8 and week 12 (follow-up visit)
Description: Overall Summary of Adverse Events is calculated on the Analysed for safety (SAF) population, i.e. 115 patients in the rhNGF group and 59 in the vehicle group.
Arm/Group | rhNGF 20 µg/ml | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/59
Serious Adverse Events (participants affected / at risk) | 1/115 | 0/59
Other Adverse Events (participants affected / at risk) | 50/115 | 19/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhNGF 20 µg/ml (N=115) | Vehicle (N=59)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.9% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhNGF 20 µg/ml (N=115) | Vehicle (N=59)
Eye pain (Eye disorders) | 23 (33) | 2 (2)
Eye irritation (Eye disorders) | 13 (21) | 10 (12)
Vision blurred (Eye disorders) | 7 (7) | 10 (12)
Myopia (Eye disorders) | 10 (10) | 4 (4)
Dry eye (Eye disorders) | 6 (8) | 6 (11)
Eye swelling (Eye disorders) | 4 (5) | 2 (2)
photophobia (Eye disorders) | 3 (4) | 3 (3)
Eyelid oedema (Eye disorders) | 3 (3) | 0 (0)
foreign body sensation in eyes (Eye disorders) | 2 (2) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 1 (2)
Diplopia (Eye disorders) | 1 (1) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 1 (1)
Ocular hyperaemia (Eye disorders) | 2 (2) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 1 (2)
Conjunctival irritation (Eye disorders) | 1 (1) | 0 (0)
Corneal epithelium defect (Eye disorders) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 9 (14) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 2 (3) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eye burns (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
LImitations and caveats non specified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT03035864/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT03035864/SAP_001.pdf